CLINICAL TRIAL: NCT06634602
Title: The Effect of Sports and Arts on Job Engagement Among Physicians: A Descriptive Study
Brief Title: The Effect of Sports and Arts on Job Engagement Among Physicians
Status: Completed | Type: Observational
Sponsor: Buğu Usanma Koban (Other)
Responsible Party: Sponsor-Investigator, Buğu Usanma Koban, Asst. Prof, Marmara University Pendik Training and Research Hospital
Organization: Marmara University Pendik Training and Research Hospital (Other)
Other Study IDs: 12.01.2024.54
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Job Engagement; Leisure Activities
Keywords: job engagement; dedication; concentration; leisure activities; healthcare professionals

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- residents, specialist physicians and academicians working in a medical faculty in İstanbul, Turkey: A survey was administered to collect sociodemographic and professional characteristics, followed by a face-to-face application of the Utrecht Work Engagement Scale (UWES-17).

SUMMARY:
The goal of this observational study was to learn about the relationship between the sociodemographic characteristics or leisure time activities of physicians and their job engagement.

The main question it aims to answer was: Do sports or artistic activities increase job engagement among physicians? A survey was administered to physicians, to collect sociodemographic and professional characteristics (including sports and artistic activities), followed by a face-to-face application of the Utrecht Work Engagement Scale (UWES-17).

ELIGIBILITY:
Inclusion Criteria:

* All physicians who agreed to participate in the study were included.

Exclusion Criteria:

* Those who did not complete the questionnaires were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All resident physicians, specialist physicians, and academic staff actively working at Marmara University School of Medicine in Istanbul.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Utrecht Work Engagement Scale (UWES-17) scores among physicians based on their engagement in sports activities | january 2024- april 2024
  Sports activities were categorized as team sports and individual sports. The frequency of activities was inquired as "I participate regularly," "I participate irregularly," or "I do not participate." Weekly activity duration was asked as "5 hours or less" and "more than 5 hours." The UWES-17 scale is compared using mean scores; there is no cut-off value, and higher scores are associated with higher job engagement.
Evaluation of the Utrecht Work Engagement Scale (UWES-17) scores among physicians based on their engagement in artistic activities | january 2024- april 2024
  Artistic activities were categorized as phonetic, rythmic and plastic art activities. The frequency of activities was inquired as "I participate regularly," "I participate irregularly," or "I do not participate." Weekly activity duration was asked as "5 hours or less" and "more than 5 hours." The UWES-17 scale is compared using mean scores; there is no cut-off value, and higher scores are associated with higher job engagement.

SECONDARY OUTCOMES:
Evaluation of the Utrecht Work Engagement Scale (UWES-17) scores among physicians based on their sociodemographic characterictics | january 2024- april 2024
  Participants' age, marital status, number of children, years spent in the medical profession, specialties, and academic titles were inquired. The responses were analyzed by comparing them with the UWES-17 scores. The UWES-17 scale is compared using mean scores; there is no cut-off value, and higher scores are associated with higher job engagement.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The participants' data will be collected online in a shared drive file.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: April 2024-June 2024
Access Criteria: being a member of research group

REFERENCES:
- [Result] Verweij H, van Hooff MLM, van der Heijden FMMA, Prins JT, Lagro-Janssen ALM, van Ravesteijn H, Speckens AEM. The relationship between work and home characteristics and work engagement in medical residents. Perspect Med Educ. 2017 Aug;6(4):227-236. doi: 10.1007/s40037-017-0364-y. PMID 28677047
- [Result] Solms L, van Vianen AEM, Theeboom T, Koen J, de Pagter APJ, de Hoog M; Challenge & Support Research Network. Keep the fire burning: a survey study on the role of personal resources for work engagement and burnout in medical residents and specialists in the Netherlands. BMJ Open. 2019 Nov 5;9(11):e031053. doi: 10.1136/bmjopen-2019-031053. PMID 31694848
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28677047/